CLINICAL TRIAL: NCT04543682
Title: A Phase I/IIa, Prospective, Mono-center, Randomized, Open Labeled, Controlled Study to Assess the Safety and Efficacy of Applying Iloprost Locally in the Fracture Site to Promote Bone Healing in Patients With Proximal Humeral Fracture
Brief Title: A Clinical Trial Investigating Iloprost as Medication to Improve Bone Healing in Patients With Proximal Humeral Fracture
Acronym: Ilobone
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Tobias Winkler, Prof. Dr. med, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIFU17; 2017-003813-24 (EudraCT Number)
Record Dates: First submitted 2020-09-02; First posted 2020-09-10 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Proximal Humeral Fracture
Keywords: proximal humeral fracture; proximale Humerusfraktur; Ilomedin; Iloprost
MeSH Terms: conditions — Shoulder Fractures | interventions — Iloprost; Open Fracture Reduction; Fracture Fixation, Internal

STUDY DESIGN:
Intervention Model Description: A randomized interventional study with parallel groups. Open labeled, add-on controlled study.
  In this study, patients will be randomized on a 1:1:1 basis to one of the three arms (two treatment arms and one control arm).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- First intervention group (0.125 ng/kg/min Iloprost) (Experimental): The first intervention group will receive open reduction and internal fixation with an angular stable plate (PHILOS™ - Depuy Synthes) + Iloprost treatment. Patients will locally receive a dose of 0.125 ng/kg/min of Iloprost over 24 hours via a catheter and an electronic pump system. The catheter will be inserted during the surgical procedure. Infusion of Iloprost will start 24hrs post-operatively and the dose will be delivered over 24h.
  Interventions: Drug: 0.125 ng/kg/min Iloprost; Procedure: open reduction and internal fixation with an angular stable plate (PHILOS)
- Second intervention group (0.25 ng/kg/min Iloprost) (Experimental): The second intervention group will also receive open reduction and internal fixation with an angular stable plate (PHILOS™ - Depuy Synthes) + Iloprost treatment. Patients will locally receive a dose of 0.25 ng/kg/min of Iloprost over 24 hours via a catheter and an electronic pump system. Infusion will start 24hrs post-operatively and the dose will be delivered over 24h.
  Interventions: Drug: 0.25 ng/kg/min Iloprost; Procedure: open reduction and internal fixation with an angular stable plate (PHILOS)
- Control intervention group (Other): Control intervention: Patients will receive the standard of care procedure for such fractures, i.e. standard of care open reduction and internal fixation with an angular stable plate (PHILOS™ - Depuy Synthes).
  Interventions: Procedure: open reduction and internal fixation with an angular stable plate (PHILOS)

INTERVENTIONS:
Drug: 0.125 ng/kg/min Iloprost — Drug administration through a catheter (inserted at the end of the surgical procedure) begins 24±2 hours after surgery: 0.125 ng/kg/min Iloprost for a duration of 24 hours
  Other Names: Ilomedin; SUB08136MIG; CAS (Chemical Abstracts Service) number 78919-13-8
  Arms: First intervention group (0.125 ng/kg/min Iloprost)
Drug: 0.25 ng/kg/min Iloprost — Drug administration through a catheter (inserted at the end of the surgical procedure) begins 24±2 hours after surgery: 0.25 ng/kg/min Iloprost for a duration of 24 hours
  Other Names: Ilomedin; SUB08136MIG; CAS number 78919-13-8
  Arms: Second intervention group (0.25 ng/kg/min Iloprost)
Procedure: open reduction and internal fixation with an angular stable plate (PHILOS) — open reduction and internal fixation with an angular stable plate (PHILOS)
  Other Names: humerus surgery; Open Reduction and Internal fixation of proximal humeral fracture using Philos plate; PHILOS Plating

SUMMARY:
The main objective of this study is to establish the safety as well as the efficacy of local insertion of Iloprost at the fracture site for bone healing of the proximal humeral fracture.

The study will have two treatment groups and one control group. All patients will receive the standard of care procedure (reduction and angular stable (PHILOS) plate fixation). The two treatment groups will additionally be treated with two different Iloprost doses.

Subjects will be assessed for study eligibility within 24h after admission (screening period). Eligible subjects will be assessed for baseline parameters on day 0. Within 96 hours of the study, subjects will undergo surgery, reduction, and angular stable (PHILOS) plate fixation. During the procedure, a catheter will be inserted in the fracture site of the treatment groups in order to deliver the Iloprost locally in the fracture site.

The expected total duration of study participation for each subject comprises 52 weeks, among which 26 weeks include active study participation. At the study end, a telephone call with the subjects will be performed for safety assessment. Recruitment will be completed in approximately 18 months.

Follow up visits following the surgical operation shall take place during weeks 3, 6, 12, and 26. The last follow-up will be a phone call during week 52 for the purpose of safety assessment.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent.
* Adult male or female subjects between 60 to 80 years old at the time of screening visit.
* Scheduled Proximal Humerus Internal Locking System (PHILOS) with 3 holes plate length for proximal humerus fracture type 3 or 4 according to Neer classification.
* Patient with American Society of Anesthesiologists (ASA) score of ≤ 2.
* Single, low energy fracture.
* Absence of neurovascular complications at the time of trauma.
* Surgery done within the first 96 hours from injury.

Exclusion Criteria:

* Subjects unable to freely give their informed consent (e.g. individuals under legal guardianship).
* Immunosuppression due to illness or medication.
* Subject with malignancy and undergoing treatment including chemotherapy, radiotherapy or immunotherapy.
* Known allergies to Iloprost.
* Conditions where the effects of Iloprost on platelets might increase the risk of haemorrhage (e.g.active peptic ulcers, or intracranial hemorrhage).
* Severe coronary heart disease or unstable angina; myocardial infarction within the last six months; decompensated cardiac failure if not under close medical supervision; severe arrhythmias; suspected pulmonary congestion; cerebrovascular events (e.g., transient ischaemic attack, stroke) within the last 3 months.
* Acute or chronic congestive heart failure (NYHA II-IV)
* Pulmonary hypertension due to venous occlusive disease.
* Congenital or acquired valvular defects with clinically relevant myocardial function disorders not related to pulmonary hypertension.
* Subject who is currently enrolled in or has not yet completed a period of at least ( a period of time equal to 5 times as the half-life time of the drug used in the previous trial) since ending other investigational device or drug trial(s).
* Patients who are dependent on the sponsor, investigator or study site.
* History of previous proximal humerus surgery on the same side.
* History of proximal humerus deformity on the same side.
* Pathological or open fracture.
* Polytrauma patient.
* Pregnant or breast-feeding women or women of childbearing potential not protected by an effective contraceptive method of birth control (defined as pearl index < 1).
* Any form of substance abuse, psychiatric disorder, or other condition that, in the opinion of the Investigator, may invalidate communication with the Investigator and/or designated study personnel.
* Patients who are committed to an institution by virtue of an order issued by either the judicial or the administrative authorities.
* Patients with a history of cerebral circulatory disorders.
* Patients with any symptomatic or treatable heart disease (including stenting), hypertension treated with a β-receptor blocker, calcium agonists, vasodilator or ACE (Angiotensin-converting-enzyme) inhibitor at more than moderate doses.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-12 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Toxicity grading in accordance with the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) | 12 months
  Toxicity grading in accordance with the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE)
Efficacy analysis using the Tip Apex Distance (TAD) readout | 12 weeks after surgery
  TAD is an indicator of the progress of fracture healing and the probability of potential complications. Thus, it reflects both the safety and efficacy of the investigational treatment. To evaluate the treatment success rate, we will calculate the percentage loss of the summation of TADs of all locking screws. The value will be classified into one of five ranks as measured after 12 weeks of postoperative follow-up compared to the baseline measurement. For the percentage of original Tip Apex Distance, the sum of the Tip Apex Distance of the humeral head screws will be used:
  Grade 1: 76%-100% preservation of the original distance (representing the best possible result), Grade 2: 51%-75% preservation of the original distance, Grade 3: 26%-50% preservation of the original distance, Grade 4: 0%-25% preservation of the original distance, and Grade 5: if the patient shows signs of screw protrusion (cut out). Grade 1 will be considered as treatment success, grades 2-5 as treatment failure.

SECONDARY OUTCOMES:
Rate of humeral head necrosis | 12 weeks and 26 weeks after surgery
  Osteonecrosis of the humeral head is a common complication in proximal humerus fracture. (1) The occurrence of osteonecrosis varies significantly according to the grading of the fracture in addition to the initial displacement (valgus or varus), Soft tissue handling during surgical fixation can influence the rate of osteonecrosis (2,3). Both a radiologist and an orthopedic surgeon will confirm the diagnosis of osteonecrosis of the humeral head radiologically at 12th-week and 26th-week visits.
Humeral head shaft angle | before discharge, 3 weeks, 6 weeks, 12 weeks and 26 weeks after surgery
  Humeral head shaft angle is used to plan corrective osteotomies and shoulder arthroplasties as well as to evaluate the postoperative x-ray outcome, as a varus displacement of more than 10 degrees in the X-ray view is considered as loss of fixation (4).
Pain assessment using the Visual Analogue Scale (VAS) | 24 hours after surgery, before discharge, 3 weeks, 6 weeks, 12 weeks and 26 weeks after surgery
  The VAS instrument consists of a 10 cm long straight line with defined endpoints, ranging from 'no pain' to 'pain as bad as it could be.' The patient will be asked to mark the respective pain level on the line that is felt subjectively. The distance between 'no pain' and the marked pain level determines the patient's pain. Scores are given in mm, ranging from 0-100 (5).
Quality-of-Life (QoL) by applying EQ-5D | 3 weeks, 6 weeks, 12 weeks and 26 weeks after surgery
  Patients will be asked to answer the questionnaire EuroQol-5 Dimension (EQ-5D), which is a validated instrument determining the quality of life as a health outcome. Developed in Europe, it is widely applied. The tool offers 5 dimensions including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression (6). The questionnaire includes a visual analog scale where patients can give information on their health state.
Constant-Murley Score (CMS): | 12 weeks and 26 weeks after surgery
  The Constant-Murley Score (CMS) is a 100-points scale composed of different parameters to define the level of pain and the ability of the patient to perform normal daily activities. It is used to determine the functional outcome after treatment of shoulder injuries. The higher the score, the better the function of the shoulder is. CMS is divided into four main subscales: pain (max. 15 points), strength (max. 25 points), daily activity (max. 20 points) and range of motion (40 points). The European Society of Shoulder and Elbow Surgery (ESSE) has promoted the Constant- Murley Score as a gold standard for the assessment of shoulder function (7-9). The Constant-Murley Score takes patient sex and age into consideration. The score can be used relative to age and sex (10).
Disabilities of the Arm, Shoulder and Hand score (DASH) | 12 weeks and 26 weeks after surgery
  DASH is a 30-item questionnaire that determines the ability of a patient to perform certain upper extremity activities. DASH questionnaire is self-reported, where patients can rate the difficulty and interference with daily life (1 = no difficulty or no symptom, 5 = unable to perform or very severe symptom). Subsequently, a score is calculated using a formula. A DASH score of 0 corresponds to no disability and 100 to extreme disability.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Winkler, Prof. Dr.med, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Center for Muskuloskeletal Surgery, Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brorson S, Rasmussen JV, Frich LH, Olsen BS, Hrobjartsson A. Benefits and harms of locking plate osteosynthesis in intraarticular (OTA Type C) fractures of the proximal humerus: a systematic review. Injury. 2012 Jul;43(7):999-1005. doi: 10.1016/j.injury.2011.08.025. Epub 2011 Oct 2. PMID 21968245
- [Background] DeFranco MJ, Brems JJ, Williams GR Jr, Iannotti JP. Evaluation and management of valgus impacted four-part proximal humerus fractures. Clin Orthop Relat Res. 2006 Jan;442:109-14. doi: 10.1097/01.blo.0000194675.64387.33. PMID 16394748
- [Background] Khmelnitskaya E, Lamont LE, Taylor SA, Lorich DG, Dines DM, Dines JS. Evaluation and management of proximal humerus fractures. Adv Orthop. 2012;2012:861598. doi: 10.1155/2012/861598. Epub 2012 Dec 18. PMID 23316376
- [Background] Malavolta EA, Assuncao JH, Pagotto RA, Avelino RL, Gracitelli ME, Pereira CA, Jacomo AL, Ferreira Neto AA. The rotation of the humeral head does not alter radiographic evaluation of the head-shaft angle. J Shoulder Elbow Surg. 2016 Apr;25(4):543-7. doi: 10.1016/j.jse.2015.09.026. Epub 2015 Dec 15. PMID 26700557
- [Background] Kersten P, White PJ, Tennant A. Is the pain visual analogue scale linear and responsive to change? An exploration using Rasch analysis. PLoS One. 2014 Jun 12;9(6):e99485. doi: 10.1371/journal.pone.0099485. eCollection 2014. PMID 24921952
- [Background] Balestroni G, Bertolotti G. [EuroQol-5D (EQ-5D): an instrument for measuring quality of life]. Monaldi Arch Chest Dis. 2012 Sep;78(3):155-9. doi: 10.4081/monaldi.2012.121. Italian. PMID 23614330
- [Background] Hirschmann MT, Wind B, Amsler F, Gross T. Reliability of shoulder abduction strength measure for the Constant-Murley score. Clin Orthop Relat Res. 2010 Jun;468(6):1565-71. doi: 10.1007/s11999-009-1007-3. Epub 2009 Jul 29. PMID 19639370
- [Background] Conboy VB, Morris RW, Kiss J, Carr AJ. An evaluation of the Constant-Murley shoulder assessment. J Bone Joint Surg Br. 1996 Mar;78(2):229-32. PMID 8666631
- [Background] Constant CR, Murley AH. A clinical method of functional assessment of the shoulder. Clin Orthop Relat Res. 1987 Jan;(214):160-4. PMID 3791738
- [Background] Yian EH, Ramappa AJ, Arneberg O, Gerber C. The Constant score in normal shoulders. J Shoulder Elbow Surg. 2005 Mar-Apr;14(2):128-33. doi: 10.1016/j.jse.2004.07.003. PMID 15789004
- [Background] Changulani M, Okonkwo U, Keswani T, Kalairajah Y. Outcome evaluation measures for wrist and hand: which one to choose? Int Orthop. 2008 Feb;32(1):1-6. doi: 10.1007/s00264-007-0368-z. Epub 2007 May 30. PMID 17534619
- [Derived] Elazaly H, Dimitriou IM, Maleitzke T, Dahne M, Jaecker V, Maerdian S, Tafelski S, Diekhoff T, Lindner T, Akgun D, Mielke AM, Paksoy A, Amini DA, Planatscher EM, Leopold V, Gonzalez-Khatib S, Kohli PC, Niemann M, Hildebrandt A, Oehme S, Palmowski Y, Paraskevaidis M, Schonnagel L, Braun SB, Pumberger M, Hardt S, Stricker S, Akyuz L, Grutz G, Schaller S, Lauterbach L, Volcksdorff M, Modl L, Textor M, Ort M, Reinke S, Stockle U, Perka C, Duda GN, Schmidt-Bleek K, Geissler S, Winkler T. ILOBONE: A phase I/IIa randomized controlled trial to assess the safety and feasibility of local iloprost therapy for enhancing proximal humerus fracture healing- a pilot study design. J Orthop Surg Res. 2025 May 22;20(1):498. doi: 10.1186/s13018-025-05865-2. PMID 40405317